CLINICAL TRIAL: NCT03630653
Title: Feasibility and Accuracy of Lymph-node (LN) Restaging by Sentinel LN Procedure and Axillary LN Dissection in Ipsilateral Invasive Breast Cancer Relapse
Brief Title: Sentinel Lymph Node Procedure in Ipsilateral Invasive Breast Cancer Relapse
Acronym: FIGARO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped prematurely due to insufficient recruitment
Sponsor: Institut Cancerologie de l'Ouest (Other)
Collaborators: Direction Générale de l'Offre de Soins (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICO-N-2017-02
Record Dates: First submitted 2018-08-07; First posted 2018-08-15 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Invasive Breast Cancer; Ipsilateral Recurrence; Sentinel Lymph Node Biopsy
Keywords: Neoplasm Staging; Neoplasm Recurrence; Axillary lymph node dissection; Conservative surgery
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sentinel LN in breast cancer recurrence (Experimental): Patients with a biopsy assessing an ipsilateral breast tumor recurrence, and a diagnosis of invasive carcinoma after a previous diagnosis of breast cancer that has been treated by breast conservative surgery at least one year before.
  Before the SLNB procedure, each patient will have a lymphoscintigraphy to evaluate axillary and extra axillary lymphatic mapping.
  Patients will be operated by breast conservative surgery (BCS) or mastectomy. Each patient will have a second SLND followed by a systematic complete ALND.
  Interventions: Procedure: Sentinel LN in breast cancer recurrence

INTERVENTIONS:
Procedure: Sentinel LN in breast cancer recurrence — Sentinel Lymph-Node (LN) procedure and Axillary LN dissection ; Mastectomy or breast conservative surgery

SUMMARY:
Sentinel lymph node biopsy (SLNB) has become the standard procedure for staging of patients with clinically node-negative breast cancer.

Breast-conserving surgery (BCS) has also been a standard treatment for patients with early breast cancer. However, approximately 10% of patients with BCS develop ipsilateral breast tumor recurrence (IBTR), and mastectomy or resection of the recurrent tumor is generally performed.

There are no specific guidelines available regarding staging and treatment of the regional lymph nodes. However, the reported risk of axillary lymph node metastasis among patients with local recurrence after breast surgery and a previous negative sentinel node biopsy of 26 % is too high to be ignored.

Moreover, evaluation of the regional lymph node basins might be helpful to decide on the indication for adjuvant radiotherapy and systemic treatment. For these reasons it seems sensible to perform a regional lymph node staging procedure in patients with locally recurrent breast cancer.

In general practice, this would mean that patients with recurrent breast cancer and a previous negative sentinel node biopsy would receive an axillary lymph node dissection (ALND) and that patients with a previous ALND would receive no additional axillary staging.

Lymphatic drainage after previous breast surgery and/or radiotherapy would be altered and it remains questionable whether SLNB at the time of surgery for IBTR (second SLNB) is technically feasible and ALND can safely be omitted.

In this study, investigators propose for all patients the realization of SLNB procedure and systematically ALND whatever the results of SLNB analysis, only on patients previously treated with breast conservative surgery.

The aim of this study is to evaluate on a homogeneous prospective multicentric cohort of patients the feasibility and the accuracy of a second SLNB procedure for IBTR.

DETAILED DESCRIPTION:
FIGARO is a prospective multicentre phase-2 study that aims to evaluate technical feasibility and validity of performing second sentinel lymph node dissection (SLND) in patients with IBTR .

To be included, patients must have a biopsy assessing an ipsilateral breast tumor recurrence, and a diagnosis of invasive carcinoma after a previous diagnosis of breast cancer that has been treated by breast conservative surgery at least one year before (time between the end of the previous radiotherapy and the diagnosis of recurrence).

At time of recurrence, the patients must be evaluated by X-ray mammography and ultrasonography examination of breast and axilla, and a full general assessment to eliminate distant metastasis.

Local recurrences will be operated by breast conservative surgery (BCS) or mastectomy. The decision between BCS and mastectomy will be carefully considered, in accordance with patient preference and other clinical features such as tumor location, tumor size, and breast size taken into account.

Each patient will have a second SLNB followed by a systematic complete ALND. Before the SLNB procedure, each patient will have a lymphoscintigraphy to evaluate axillary and extra axillary lymphatic mapping. Lymphoscintigraphy will be performed according to previously reported standard techniques. At 2-20 h after lymphoscintigraphy, SLNB will be performed with or without a blue dye associated injection. An intraoperative gamma ray detection probe will be used during surgery to conﬁrm locations of the sentinel nodes and to facilitate their removal. All sentinel nodes will be removed and sent for histopathologic examination according to previously described standard techniques. A complete ALND (Berg's stage I and II) will be realized and the nodes will be sent for standard histopathologic examination.

Further systemic adjuvant therapies will be chosen in a multidisciplinary approach considering prognostic and predictive indicators.

All the patients will be followed up for 5 years at 12-month intervals after the second surgery and undergo annual mammography with or without ultrasonography.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years old
2. Invasive recurrence (ductal, lobular, other), homolateral breast carcinoma
3. Size of the tumor with ultrasound ≤ 5cm
4. Initial conservative surgery
5. Patient who has already received SLND for her initial cancer, regardless of the SLND result
6. Procedure for the detection of lymph node sentinel by isotopic method +/- colorimetric
7. Minimum delay of one year between the end of radiotherapy for initial breast carcinoma and the treatment / management of ipsilateral recurrence
8. Pregnancy test (urinary or blood) negative for premenopausal patients
9. Information of the patient and obtaining written consent, signed by the patient and the investigator

Exclusion Criteria:

1. Non-invasive recurrence
2. History of ipsilateral axillary dissection
3. History of ipsilateral mastectomy
4. Patient pN + before surgery
5. Metastasis
6. Allergy known to 2 detection products (Blue and radioactive tracer)
7. Pregnant or lactating woman
8. Patient protected or under guardianship or unable to give consent
9. Impossibility of submitting to the medical examination for geographical, social or psychological reasons

Min Age: 18 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2020-12-03 (Actual); Study Completion 2020-12-03 (Actual)

PRIMARY OUTCOMES:
False-negative rate in patients with a second SLNB procedure for IBTR | 30 days post-surgery
  Ratio of the number of cases with detection of negative sentinel axillary lymph node but with at least one metastatic lymph node in the axillary dissection on the total number of patients with at least one detected a sentinel axillary node and at least one metastatic lymph node, either in a sentinel axillary lymph node or in complete ALND

SECONDARY OUTCOMES:
Detection rate | 1 to 2 hours post-surgery
  Ratio of the number of patients injected, technetium +/- blue, in which at least one sentinel axillary lymph node was detected intraoperative on the total number of patients injected
lymph node involvement | 30 days post-surgery
  % of lymph node involvement
patient requiring consolidation radiotherapy | 30 days post-surgery
  % of patient requiring consolidation radiotherapy on axillary and extra-axillary lymph node sites
% of extra-axillary positivity by lymphoscintigraphy | Within 24 hours before surgery
  Lymphoscintigraphy will be performed within 24 hours before surgery
Recurrence Free Survival (RFS) | Up to 5 years post-surgery
  Time until recurrence

CONTACTS AND LOCATIONS:
Overall Officials: VIRGINIE BORDES, MD, Study Director — ICO
Locations (9):
- France (9):
  - Institut Bergonie, Bordeaux
  - CENTRE REGIONAL DE LUTTE CONTRE LE CANCER D'AUVERGNE - centre JEAN PERRIN, Clermont-Ferrand
  - Centre Georges Francoise Leclerc, Dijon
  - ICM Val d'Aurelle, Montpellier
  - INSTITUT REGIONAL DU CANCER MONTPELLIER - Val D'Aurelle, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Saint-Cloud
  - Ico Nantes, Saint-Herblain
  - IUCT-O Institut Claudius Regaud, Toulouse

IPD SHARING:
Plan to Share IPD: No